CLINICAL TRIAL: NCT03773289
Title: Drug Utilization Patterns in Neonatal Units in the UK: a Retrospective Pharmaco-epidemiological Study
Brief Title: Commonly Used Medicines On Neonatal Units in the UK
Acronym: COMMON
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 18023
Record Dates: First submitted 2018-12-05; First posted 2018-12-12 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2020-03

CONDITIONS: Infant, Newborn; Pharmacoepidemiology; Intensive Care Units, Neonatal
Keywords: Infants, neonates; rational drug use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is a retrospective, observational pharmacoepidemiological study using nationally collected data. There is no intervention.

SUMMARY:
This retrospective analysis of drug utilisation data aims to study the patterns of use of medicines in neonatal units in the UK from 2010 to 2017. Prescribing drugs in neonates can be complex and the application of pharmacotherapy principles can be challenging due to the lack of licenced formulations and limited evidence-base for indications, dosing and/or adverse events. A systematic review of drug utilisation pattern in neonatal units in different health care settings identified antibiotics, caffeine and vitamin supplements as the most commonly used drugs and highlighted that further research is needed to investigate drug utilisation and rational use of medicines in neonates. The only UK study included in this systematic review and available from our search of literature was conducted in 2009. This survey, however, had a low response rate (only 42% units responded) and it included data collection over a very short period of 2 weeks and that could limit its generalisability to other NICU settings. It identified the need for research in to medicines for neonates and that this research agenda should be informed by the extent of medication use in this field. However, our literature search revealed that there is very little information on the current patterns of medication use in neonates. An updated drug utilisation study is warranted in a neonatal setting in UK.

DETAILED DESCRIPTION:
The aim of this study is to investigate current and recent patterns of drug utilisation in neonatal units in the UK.

We will conduct a retrospective pharmacoepidemiological study of a large prospectively collected database (The National Neonatal Research Database -REC Number 16/LO/1093). The study will use de-identified historical data recorded in this database. There is no patient recruitment and the project involves no changes to patient care. The data to be used for this project are stored in de-identified form.

Data items will include descriptive, background data to allow for age and gestation at the time of drug use and subgroup analysis (such as birth weight, gestational age, clinical condition, day of drug use) and data on drug use (name of drug and age at use).

ELIGIBILITY:
Inclusion criteria

* Infants admitted to neonatal units in England, Scotland, and Wales
* Admitted between 01 January 2010 and 31 December 2017.
* No limits in gestational age or birth weight.

Exclusion cirteria

* Infants who received all their care in the postnatal ward
* Infants who were not admitted to any neonatal unit

Ages: 0 Weeks to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Inclusion criteria
  * Infants admitted to neonatal units in England, Scotland, and Wales
  * Admitted between 01 January 2010 and 31 December 2017.
  * No limits in gestational age or birth weight.
  Exclusion cirteria
  * Infants who received all their care in the postnatal ward
  * Infants who were not admitted to any neonatal unit
Sampling Method: Non-Probability Sample
Enrollment: 642729 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2020-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Most commonly prescribed drugs in neonatal units in the UK | Last 8 years [01/01/2010 -31/12/2017]
  List the most commonly prescribed drugs in neonatal units in the UK (proportion of all infants exposed to each drug at least once during their admission)
Change in pattern of drug use over 8 years in the UK | Last 8 years [01/01/2010 -31/12/2017]
  listing the most frequently used drugs by year.

SECONDARY OUTCOMES:
List of the most frequently used drugs by gestation category | Last 8 years [01/01/2010 -31/12/2017]
  gestational category according to WHO definition (term: more than or equal to 37 weeks, moderate to late 32-36 weeks, very preterm 28-31 weeks, extremely preterm < 28 weeks)
Figures for the average duration of drug exposure by gestation category | Last 8 years [01/01/2010 -31/12/2017]
  gestational category according to WHO definition[term: more than or equal to 37 weeks, moderate to late 32-36 weeks, very preterm 28-31 weeks, extremely preterm < 28 weeks]
List of the most frequently used drugs by care level of admitting neonatal unit | Last 8 years [01/01/2010 -31/12/2017]
  The definition is (Level 3 Neonatal Intensive Care Units; Level 2 Local Neonatal Units)
Figures for the average duration of drug exposure by birth weight | Last 8 years [01/01/2010 -31/12/2017]
  The birth weight is grouped in 250g increments from <500g to >2500g

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Ojha, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Division of Graduate Entry Medicine-School of Medicine, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Turkait A, Szatkowski L, Choonara I, Ojha S. Management of patent ductus arteriosus in very preterm infants in England and Wales: a retrospective cohort study. BMJ Paediatr Open. 2022 Mar;6(1):e001424. doi: 10.1136/bmjpo-2022-001424. PMID 36053632
- [Derived] Al-Turkait A, Szatkowski L, Choonara I, Ojha S. Drug utilisation in neonatal units in England and Wales: a national cohort study. Eur J Clin Pharmacol. 2022 Apr;78(4):669-677. doi: 10.1007/s00228-021-03267-x. Epub 2022 Jan 13. PMID 35028673